CLINICAL TRIAL: NCT06482632
Title: The Effect of the Transection of the Omohyoid in the Incidence of Dysphagia in Patients Undergoing Multilevel Anterior Cervical Discectomy and Fusion
Brief Title: The Effect of the Transection of the Omohyoid in the Incidence of Dysphagia in Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 119384
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Anterior Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: This study intends to report the incidence of dysphagia in patients who underwent multilevel Anterior Cervical Discectomy and Fusion with or without omohyoid transection during the surgical approach. Patients selected for this study will be those who are treated at the University District Hospital (UDH) of the UPR - SOM.
  The study is composed of patients who underwent ACDF at our institutions. Randomization of dissected Omohyoid was performed utilizing an online computer-generated sequence (www.graphpad.com/quickcalcs/randomN1.cfm). A request for the waiver of authorization to release health information will be completed. After the research committee approves, medical records will be reviewed to gather information such as age, gender, smoking status, diabetic status, body mass index (BMI), inpatient medications, and discharge medications. After discharge, patients undergoing this procedure are followed up at outpatient clinics.
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discectomy of Omohyoid (Other): Patient undergoing an anterior cervical discectomy (ACDF) and fusion will have the Omohyoid removed to determine the effect of dysphagia after surgery.
  Interventions: Procedure: Discectomy of Omohyoid
- No discectomy of Omohyoid (Other): Patient undergoing an anterior cervical discectomy (ACDF) and fusion will not have the Omohyoid removed to determine the effect of dysphagia after surgery.
  Interventions: Procedure: Control group no discectomy of Omohyoid

INTERVENTIONS:
Procedure: Discectomy of Omohyoid — Will be removing the Omohyoid during an anterior cervical discectomy and fusion to compare its effect of dysphagia.
  Arms: Discectomy of Omohyoid
Procedure: Control group no discectomy of Omohyoid — Will not be removing the Omohyoid during an anterior cervical discectomy and fusion to compare its effect of dysphagia.
  Arms: No discectomy of Omohyoid

SUMMARY:
The investigators believe that the transection of the omohyoid during an anterior cervical discectomy and fusion decreases the incidence of dysphagia in patients who undergo this procedure when compared to patients who do not have the omohyoid transected.

DETAILED DESCRIPTION:
Dysphagia is a common postoperative complication in patients undergoing anterior cervical discectomy and fusion (ACDF). Although it is often transient, there have been cases of postoperative dysphagia lasting for several months or being permanent. The pathogenesis of this complication is poorly understood and likely multifactorial. There have been multiple risk factors described that may contribute to postoperative dysphagia, but there is a lack of clarity regarding these. The effect of transecting the omohyoid during a multilevel Anterior Cervical Discectomy and Fusion has been controversial. The transaction of this muscle is generally safe and is often used during the approach of the technique for improved visualization.

This research study aims to determine whether the transection of the omohyoid affects the incidence of dysphagia in patients who underwent multilevel ACDF and whether it should be routinely performed during a multilevel ACDF. The investigators plan to prospectively enroll 60 patients undergoing multilevel ACDF (C3-C7). Patients selected in the allotted time frame were treated by the orthopedic spine service of the University of Puerto Rico Orthopaedic Surgery Residency Program. Exclusion criteria include those patients with preoperative dysphagia, those with conditions that expose them to a high risk of postoperative dysphagia (such as motor neuron disease), and those with cervical non-degenerative pathology, such as tumor or trauma. Randomization was performed utilizing an online computer-generated sequence (www.graphpad.com/quickcalcs/randomN1.cfm). A request for the waiver of authorization to release health information will be completed. After the research committee approves, medical records will be reviewed to gather information such as age, gender, smoking status, diabetic status, body mass index (BMI), inpatient medications, and discharge medications. After discharge, patients undergoing this procedure are followed up at outpatient clinics (Clinicas Externas). Follow-up intervals include postoperative days 1 and 2, 4, and 8 weeks after surgical intervention. On the first postoperative day, and each of the follow-up visits we will collect dysphagia scores via a modified Swallowing Quality of Life Scale (Swal-QOL) and physician notes. Physician notes will also be evaluated for clear documentation of patient-reported outcomes. Results will be gathered to evaluate outcomes and complications.

The target population is female and male patients between 21 - 85 years old undergoing multilevel anterior cervical decompression and fusion.

Patients with a history of preoperative dysphagia, those with conditions that expose them to high risk of postoperative dysphagia (such as motor neuron disease), and those with cervical non-degenerative pathology, such as tumor or trauma as well as those who have lost to follow up, will be excluded from the study.

The risks of participating in this study, though minimal, include a breach in confidentiality. The benefits of participation include contributing to the Orthopaedic Surgery research community to guide future pain management in fracture care.

To ensure the confidentiality of subjects' data, all information gathered from medical records (MR) will be de-identified and stored in a password-protected database. The database will only be accessible to Principal Investigators, CO-Principal Investigators, and students from the Orthopaedic Surgery Department, who meet all "CITI Program" requirements and have completed HIPAA training. An identification number will be assigned to each participant to not use the patient's number from the Medical Record. Data for age, gender, smoking status, diabetic status, body mass index (BMI), inpatient medications, and discharge medications will be collected apart from Medical Record numbers and identifiable data. These documents can only be accessed by those electronically permitted by the Principal Investigator, furthermore, a unique password has to be written, to access the database. Therefore, since there are different measures to ensure privacy (electronic permit granted by Principal Investigator and password protection), we understand that this research ensures adequate parameters for confidentiality. After data collection and statistical analysis are done, the password-protected database will be made inaccessible, deleted, and destroyed to preclude reproduction and divulgation of data. Identifiers will not be maintained following the completion of the study. The study is composed of patients who underwent Principal Investigators at our institutions. The sub-groups will be created based on the transaction of omohyoid (transected vs non-transected) to allow comparisons in Sociodemographic information, past medical history, body mass index and confounding variables that might affect our results are: patient comorbidities, gender, and levels of fused. Finally the population selected may represent convenience bias due to its location on the northeast side of Puerto Rico.

ELIGIBILITY:
Inclusion Criteria:

* The target population is female and male patients between 21 - 85 years old undergoing multilevel anterior cervical decompression and fusion.

Exclusion Criteria:

* Patients with a history of preoperative dysphagia, those with conditions that expose them to high risk of postoperative dysphagia (such as motor neuron disease), and those with cervical non-degenerative pathology, such as tumor or trauma as well as those who have lost to follow up, will be excluded from the study.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 6 months
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.
Dysphagia Short Questionnaire- "The Dysphagia Questionnaire | 6 months
  a 10-point rating scale, were 1 is the minimum value, 10 is the maximum value, and the higher scores means the worse outcome and lower scores are the better outcomes. In the Dysphagia questionnaire the patients provide an assessment of the severity of dysphagia symptoms experienced.

SECONDARY OUTCOMES:
Neck Circumference | Pre operation
  Measurement of neck circumference in centimeters
Body Mass Index | Pre Operation
  Measure the body mass index of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Oncológico Dr. Isaac González Martínez, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No